CLINICAL TRIAL: NCT07263516
Title: Effects of Combined Pelvic Floor and Diaphragmatic Breathing Exercises on Primary Dysmenorrhea
Brief Title: Pelvic Floor and Diaphragmatic Breathing Exercises for Primary Dysmenorrhea
Acronym: PFDD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Irmak KARDEŞ, Graduate Student, Istanbul Gelisim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulGelisimU-FTR-IK-01
Record Dates: First submitted 2025-09-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Primary Dysmenorrhea (PD)
Keywords: primary dysmenorrhea; Menstrual pain; Pelvic floor exercises; Diaphragmatic breathing; Physiotherapy; Pain management; Exercise therapy; Biopsychosocial model; Depression, anxiety, stress; Sleep quality; Non-pharmacological treatment; Randomized controlled trial (RCT); Women's health
MeSH Terms: conditions — Dysmenorrhea; Agnosia; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two parallel groups. The intervention group will perform a combined program of pelvic floor muscle and diaphragmatic breathing exercises, while the control group will perform only diaphragmatic breathing exercises. Both groups will be assessed at two time points: before and after the menstrual period.
Masking Description: This is an open-label study. No participants, care providers, investigators, or outcome assessors are blinded to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intervention group → Pelvic floor + diaphragmatic breathing exercises (Experimental): Participants will perform a combined program of pelvic floor muscle exercises and diaphragmatic breathing exercises. The exercises will be conducted according to the study protocol, with sessions scheduled regularly over the intervention period. Both physical and psychological outcomes will be assessed before and after the menstrual period.
  Interventions: Behavioral: Pelvic Floor + Breathing Exercises
- Arm 2: Control group: Diaphragmatic breathing exercises (Active Comparator): Participants will perform only diaphragmatic breathing exercises according to the study protocol. Assessments of pain, menstrual symptoms, quality of life, sleep quality, and psychological measures will be conducted before and after the menstrual period.
  Interventions: Behavioral: Diaphragmatic Breathing Exercises

INTERVENTIONS:
Behavioral: Pelvic Floor + Breathing Exercises — Participants will perform both pelvic floor and diaphragmatic breathing exercises according to the study protocol. Assessments will focus on pain, quality of life, and psychological measures.
  Arms: Arm 1: Intervention group → Pelvic floor + diaphragmatic breathing exercises
Behavioral: Diaphragmatic Breathing Exercises — Participants will perform only diaphragmatic breathing exercises. Assessments will be conducted in the same manner.
  Arms: Arm 2: Control group: Diaphragmatic breathing exercises

SUMMARY:
This study investigates whether combining pelvic floor muscle exercises with diaphragmatic breathing exercises can reduce menstrual pain in women with primary dysmenorrhea. Forty participants will be randomly assigned to two groups: one performing both exercises, and the other performing only diaphragmatic breathing. The study will measure pain, menstrual symptoms, quality of life, and psychological well-being before and after the intervention.

DETAILED DESCRIPTION:
This interventional study aims to investigate the combined effects of pelvic floor muscle exercises and diaphragmatic breathing exercises on primary dysmenorrhea in women. The study is designed based on a biopsychosocial model to explore both physical and psychological outcomes of the intervention.

A total of 40 participants will be recruited and randomly assigned to two groups. The intervention group will perform a program combining pelvic floor and diaphragmatic breathing exercises, while the control group will perform only diaphragmatic breathing exercises. The exercise program will be conducted over a specified period, with sessions scheduled regularly according to the study protocol.

Assessments will be conducted twice: prior to and after the menstrual period. Pain intensity will be evaluated using the Visual Analog Scale (VAS), and pain threshold will be measured with a pressure algometer. Menstrual and premenstrual symptoms, quality of life, sleep quality, and psychological status, including depression, anxiety, and stress levels, will be assessed using validated scales such as the PMS Scale, SF-36, DASS-21, and PUKI.

This study is expected to provide scientific evidence for physiotherapy interventions in women's health and offer an alternative non-pharmacological approach for managing primary dysmenorrhea. By addressing both physical and psychological aspects, the exercise program may reduce pain, improve quality of life, and enhance overall well-being in participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Diagnosed with primary dysmenorrhea (PD)
* Having regular menstrual cycles for the past 6 months
* Willing to participate in the study

Exclusion Criteria:

* Diagnosis of secondary dysmenorrhea
* Irregular menstrual cycles (less than 21 days or more than 35 days)
* History of childbirth or previous pregnancy
* Currently pregnant
* Presence of any neurological, systemic, or psychiatric chronic disease
* Regular use of medications in the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who identify as female and have a uterus are eligible to participate.
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (Visual Analog Scale, VAS) | 1-2 days before the onset of menstruation (pre-menstrual assessment) and 1-2 days after the end of menstruation (post-menstrual assessment).
  Pain severity will be assessed using a 100-mm Visual Analog Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Participants will mark their perceived pain level, which will then be measured with a ruler to obtain a numerical value.
Pain Threshold (Pressure Algometer) | 1-2 days before the onset of menstruation (pre-menstrual assessment) and 1-2 days after the end of menstruation (post-menstrual assessment).
  Pain threshold will be assessed at six anatomical points using a pressure algometer. Pressure is gradually increased until participants report pain. Two measurements per point are recorded, with the mean value calculated in lbs/cm².
Menstrual Symptoms (Menstrual Symptom Scale - MSS) | 1-2 days before the onset of menstruation (pre-menstrual assessment) and 1-2 days after the end of menstruation (post-menstrual assessment).
  The severity of menstrual symptoms will be assessed using the Menstrual Symptom Scale (MSS), whose Turkish validity and reliability were established by Güvenç, Seven, and Akyüz (2014). The scale consists of 22 items, each rated on a 5-point Likert scale from 1 ("never") to 5 ("always").
  Minimum possible total score: 22 points Maximum possible total score: 110 points
Premenstrual Symptoms (PMS Scale) | One week before menstruation
  Premenstrual symptoms will be assessed using the 44-item PMS Scale, covering nine subscales such as depressive mood, anxiety, fatigue, irritability, pain, sleep, and appetite changes. The total score of the scale is obtained by summing the scores from all subscales, ranging from 44 to 220 points. Higher scores indicate a greater severity of premenstrual syndrome (PMS) symptoms.

SECONDARY OUTCOMES:
Quality of Life (SF-36) | 1-2 days before the onset of menstruation (pre-menstrual assessment) and 1-2 days after the end of menstruation (post-menstrual assessment).
  The Short Form-36 (SF-36) questionnaire evaluates physical and mental health across 8 subscales. Scores range from 0-100, with higher scores indicating better quality of life.
Sleep Quality (Pittsburgh Sleep Quality Index - PSQI) | 1-2 days before the onset of menstruation (pre-menstrual assessment) and 1-2 days after the end of menstruation (post-menstrual assessment).
  Sleep quality will be measured with the PSQI, a 24-item questionnaire assessing sleep duration, quality, disturbances, and daytime dysfunction. Total scores range from 0-21; higher scores indicate poorer sleep quality.
Depression, Anxiety, and Stress (DASS-21) | 1-2 days before the onset of menstruation (pre-menstrual assessment) and 1-2 days after the end of menstruation (post-menstrual assessment).
  DASS-21 assesses levels of depression, anxiety, and stress across 21 items. Each subscale includes 7 items, rated on a 0-3 Likert scale. Higher scores indicate greater severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Irmak KARDEŞ, Principal Investigator — Istanbul Gelişim University
Locations (1):
- Istanbul Gelişim University, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dixon JS, Bird HA. Reproducibility along a 10 cm vertical visual analogue scale. Ann Rheum Dis. 1981 Feb;40(1):87-9. doi: 10.1136/ard.40.1.87. PMID 7469530
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Brown TA, Chorpita BF, Korotitsch W, Barlow DH. Psychometric properties of the Depression Anxiety Stress Scales (DASS) in clinical samples. Behav Res Ther. 1997 Jan;35(1):79-89. doi: 10.1016/s0005-7967(96)00068-x. PMID 9009048
- [Result] ACOG Committee Opinion No. 760: Dysmenorrhea and Endometriosis in the Adolescent. Obstet Gynecol. 2018 Dec;132(6):e249-e258. doi: 10.1097/AOG.0000000000002978. PMID 30461694